CLINICAL TRIAL: NCT06991231
Title: The Benefits Of Cryoablation In Patients Undergoing Total Knee Arthroplasty - A Randomized Prospective Clinical Trial
Brief Title: The Benefits Of Cryoablation In Patients Undergoing Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-00306
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-05-27 (Actual); Status verified 2025-05

CONDITIONS: Post-Operative Pain; Total Knee Arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Arthroplasty, Replacement, Knee; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Total knee arthroplasty (TKA) + Cryoablation (Experimental): Patients will receive cryoablation during the two to three weeks prior to the TKA procedure.
  Interventions: Procedure: Total knee arthroplasty (TKA); Device: Cryoablation
- TKA Only (Active Comparator): Patients will NOT receive cryoablation prior to the TKA procedure.
  Interventions: Procedure: Total knee arthroplasty (TKA)

INTERVENTIONS:
Procedure: Total knee arthroplasty (TKA) — Administered as part of patient standard of care.
Device: Cryoablation — Cryoablation will be administered on the leg of the knee indicated for surgery.
  Arms: Total knee arthroplasty (TKA) + Cryoablation

SUMMARY:
The purpose of this study is to evaluate the efficacy of cryoablation use on patient-reported outcomes (PROMs) and opioid consumption following total knee arthroplasty. This is a randomized study that will involve a 1:1 randomization to total knee arthroplasty +/- cryoablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients are candidates for elective primary total knee arthroplasty for a diagnosis of osteoarthritis or inflammatory arthritis.
* Patients have been medically cleared and scheduled for surgery

Exclusion Criteria:

* Patients with cold-related conditions (cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, and Raynaud's disease)
* Surgery for fracture, infection, or malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption during Post-Procedural Follow-Up Period | Month 3 Post-Operation (Approximately Week 8-9)
  Measured as morphine milligram equivalents.
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) Score | Month 3 Post-Operation (Approximately Week 8-9)
  KOOS, JR. is a 7-item assessment of how participants feel about their knee and how well they are able to do usual activities. Each item is rated on a Likert scale; the raw score is the sum of item responses. The raw score is transformed into a total score ranging from 0-100, where 0 indicates total knee disability and 100 represents perfect knee health.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rozell, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Daniel.waren@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Daniel.waren@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.